CLINICAL TRIAL: NCT00429429
Title: Immunotherapy for Peanut Allergy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Wesley Burks, MD, Chairman, Department of Pediatrics, University of North Carolina, Chapel Hill
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R21AT002557-02 (NIH)
Record Dates: First submitted 2007-01-30; First posted 2007-01-31 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Allergy
Keywords: Peanut allergy
MeSH Terms: conditions — Hypersensitivity; Peanut Hypersensitivity | interventions — Sublingual Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Peanut protein solution (Experimental): Subjects receiving the peanut sublingual peanut protein drops. Sublingual Immunotherapy.
  Interventions: Procedure: Sublingual immunotherapy

INTERVENTIONS:
Procedure: Sublingual immunotherapy — Drops of peanut protein placed and held under the tongue for a specific time before swallowed.
  Other Names: Peanut protein solution

SUMMARY:
Currently, when a food allergy is diagnosed, the "standard of care" is strict avoidance of the allergic food and ready access to self-injectable epinephrine. Yet, accidental ingestions do occur. Unfortunately, for a ubiquitous food such as peanut, the possibility of an inadvertent ingestion is great. It is estimated that over 50% of individuals who are allergic to peanuts will have an accidental reaction to peanuts over a 2-year period. The purpose of this study is to determine if peanut sublingual immunotherapy (SLIT) reduces the number and/or symptoms of accidental peanut ingestion in peanut allergic subjects. We would anticipate that the subjects on the peanut SLIT protocol would experience few adverse effects with accidental peanut ingestion over the course of the two years of SLIT. The primary endpoint to evaluate the effectiveness of SLIT will be a negative DBPCFC to peanuts (8 grams) at the completion of the two years of the study.

DETAILED DESCRIPTION:
Peanut allergy is one of the most serious of the immediate hypersensitivity reactions to foods in terms of persistence and severity of the reaction and appears to be a growing problem. Allergen-specific immunotherapy (IT) is currently being examined as a treatment option because of the persistence of this hypersensitivity reaction and the lack of effective treatment. An understanding of the molecular mechanisms of peanut-specific IT is vital to ensure the eventual, successful treatment of peanut-allergic patients.

The goal of this proposal is to develop peanut immunotherapy (IT) for patients with peanut allergic reactions. This innovative application is designed to utilize the extensive knowledge of the allergens involved in peanut hypersensitivity to devise an immunotherapeutic approach that would lower the risk of anaphylactic reactions and would down regulate peanut-specific T cells in peanut-allergic patients. Previous attempts to utilize peanut-specific immunotherapy have been unsuccessful primarily because of the severe side effects of therapy.

The specific aim of the study is to desensitize/tolerize peanut-allergic subjects with peanut allergen-specific, sublingual immunotherapy (SLIT) and begin to determine the molecular mechanism of the peanut-specific T-cell response during SLIT.

The hypothesis is that peanut SLIT will desensitize patients with peanut allergic reactions by the induction of peanut specific regulatory T cells resulting in immune modulation of the peanut allergic reaction.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 6 and 35 years of age
* Diagnosed with peanut allergy by positive prick skin test, CAP FEIA of 15 Ku/L or greater
* History of significant clinical symptoms within one hour after ingestion of peanuts
* Family's compliance with all study visits

Exclusion Criteria:

* Subjects with medical history preventing a BDPCFC to peanut
* Subjects unable to cooperate with challenge procedure
* Subjects unable to be reached by telephone for follow-up
* Subjects with a history of severe anaphylaxis to peanut

Ages: 6 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2006-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
A negative double-blind placebo controlled food challenge at the completion the two years of the study. | When IgE level drops to less than or equal to 2 ku/L

SECONDARY OUTCOMES:
A change in the cytokine level between the baseline and each selected time point during the two years of the study. | Drop in cytokine level

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Burks, MD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bock SA, Munoz-Furlong A, Sampson HA. Fatalities due to anaphylactic reactions to foods. J Allergy Clin Immunol. 2001 Jan;107(1):191-3. doi: 10.1067/mai.2001.112031. PMID 11150011
- [Background] Sicherer SH, Munoz-Furlong A, Burks AW, Sampson HA. Prevalence of peanut and tree nut allergy in the US determined by a random digit dial telephone survey. J Allergy Clin Immunol. 1999 Apr;103(4):559-62. doi: 10.1016/s0091-6749(99)70224-1. PMID 10200001
- [Background] Sicherer SH, Munoz-Furlong A, Sampson HA. Prevalence of peanut and tree nut allergy in the United States determined by means of a random digit dial telephone survey: a 5-year follow-up study. J Allergy Clin Immunol. 2003 Dec;112(6):1203-7. doi: 10.1016/s0091-6749(03)02026-8. PMID 14657884
- [Background] Oppenheimer JJ, Nelson HS, Bock SA, Christensen F, Leung DY. Treatment of peanut allergy with rush immunotherapy. J Allergy Clin Immunol. 1992 Aug;90(2):256-62. doi: 10.1016/0091-6749(92)90080-l. PMID 1500630
- [Background] Wilson DR, Torres LI, Durham SR. Sublingual immunotherapy for allergic rhinitis. Cochrane Database Syst Rev. 2003;(2):CD002893. doi: 10.1002/14651858.CD002893. PMID 12804442
- [Background] Sloan AE, Powers ME. A perspective on popular perceptions of adverse reactions to foods. J Allergy Clin Immunol. 1986 Jul;78(1 Pt 2):127-33. doi: 10.1016/0091-6749(86)90002-3. No abstract available. PMID 3722639
- [Background] Jansen JJ, Kardinaal AF, Huijbers G, Vlieg-Boerstra BJ, Martens BP, Ockhuizen T. Prevalence of food allergy and intolerance in the adult Dutch population. J Allergy Clin Immunol. 1994 Feb;93(2):446-56. doi: 10.1016/0091-6749(94)90353-0. PMID 8120272
- [Background] Sampson HA. Food allergy. J Allergy Clin Immunol. 1989 Dec;84(6 Pt 2):1062-7. doi: 10.1016/0091-6749(89)90154-1. No abstract available. PMID 2600342
- [Background] Bock SA, Atkins FM. Patterns of food hypersensitivity during sixteen years of double-blind, placebo-controlled food challenges. J Pediatr. 1990 Oct;117(4):561-7. doi: 10.1016/s0022-3476(05)80689-4. PMID 2213379
- [Background] Valentine MD, Schuberth KC, Kagey-Sobotka A, Graft DF, Kwiterovich KA, Szklo M, Lichtenstein LM. The value of immunotherapy with venom in children with allergy to insect stings. N Engl J Med. 1990 Dec 6;323(23):1601-3. doi: 10.1056/NEJM199012063232305. PMID 2098016
- [Background] Leung DY, Sampson HA, Yunginger JW, Burks AW Jr, Schneider LC, Wortel CH, Davis FM, Hyun JD, Shanahan WR Jr; Avon Longitudinal Study of Parents and Children Study Team. Effect of anti-IgE therapy in patients with peanut allergy. N Engl J Med. 2003 Mar 13;348(11):986-93. doi: 10.1056/NEJMoa022613. Epub 2003 Mar 10. PMID 12637608
- [Background] Scadding GK, Brostoff J. Low dose sublingual therapy in patients with allergic rhinitis due to house dust mite. Clin Allergy. 1986 Sep;16(5):483-91. doi: 10.1111/j.1365-2222.1986.tb01983.x. PMID 3536171
- [Background] Tonnel AB, Scherpereel A, Douay B, Mellin B, Leprince D, Goldstein N, Delecluse P, Andre C. Allergic rhinitis due to house dust mites: evaluation of the efficacy of specific sublingual immunotherapy. Allergy. 2004 May;59(5):491-7. doi: 10.1111/j.1398-9995.2004.00456.x. PMID 15080829
- [Background] Canonica GW, Passalacqua G. Noninjection routes for immunotherapy. J Allergy Clin Immunol. 2003 Mar;111(3):437-48; quiz 449. doi: 10.1067/mai.2003.129. PMID 12642818
- [Background] Morris DL. Treatment of respiratory disease with ultra-small doses of antigens. Ann Allergy. 1970 Oct;28(10):494-500. No abstract available. PMID 5521180
- [Background] Holt PG, Sly PD, Smith W. Sublingual immunotherapy for allergic respiratory disease. Lancet. 1998 Feb 28;351(9103):613-4. doi: 10.1016/S0140-6736(05)78425-7. No abstract available. PMID 9500315
- [Background] Grosclaude M, Bouillot P, Alt R, Leynadier F, Scheinmann P, Rufin P, Basset D, Fadel R, Andre C. Safety of various dosage regimens during induction of sublingual immunotherapy. A preliminary study. Int Arch Allergy Immunol. 2002 Nov;129(3):248-53. doi: 10.1159/000066779. PMID 12444323
- [Background] Bousquet J, Michel FB. Specific immunotherapy in asthma. Allergy Proc. 1994 Nov-Dec;15(6):329-33. doi: 10.2500/108854194778816562. PMID 7721083
- [Background] Morris DL, Kroker GF, Sabnis VK, Morris MS. Local immunotherapy in allergy. Chem Immunol Allergy. 2003;82:1-10. doi: 10.1159/000071537. PMID 12947987
- [Background] Taams LS, Vukmanovic-Stejic M, Smith J, Dunne PJ, Fletcher JM, Plunkett FJ, Ebeling SB, Lombardi G, Rustin MH, Bijlsma JW, Lafeber FP, Salmon M, Akbar AN. Antigen-specific T cell suppression by human CD4+CD25+ regulatory T cells. Eur J Immunol. 2002 Jun;32(6):1621-30. doi: 10.1002/1521-4141(200206)32:63.0.CO;2-Q. PMID 12115645
- [Background] Li XM, Serebrisky D, Lee SY, Huang CK, Bardina L, Schofield BH, Stanley JS, Burks AW, Bannon GA, Sampson HA. A murine model of peanut anaphylaxis: T- and B-cell responses to a major peanut allergen mimic human responses. J Allergy Clin Immunol. 2000 Jul;106(1 Pt 1):150-8. doi: 10.1067/mai.2000.107395. PMID 10887318
- [Background] Lee SY, Huang CK, Zhang TF, Schofield BH, Burks AW, Bannon GA, Sampson HA, Li XM. Oral administration of IL-12 suppresses anaphylactic reactions in a murine model of peanut hypersensitivity. Clin Immunol. 2001 Nov;101(2):220-8. doi: 10.1006/clim.2001.5122. PMID 11683581
- [Background] Cohen J. Statistical power analysis for the behavioral sciences. 2nd edition ed. Hillsdale, NJ: Erlbaum, 1988.